CLINICAL TRIAL: NCT00973778
Title: A Phase II Study for Short Preoperative Chemoradiotherapy Utilizing Intensity Modulated Radiation Therapy (IMRT) in Combination With Capecitabine in Patients With Resectable Rectal Carcinoma
Brief Title: A Study for Short Preoperative Chemoradiotherapy for Resectable Rectal Carcinoma
Acronym: IMRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Weiguo Cao, Shanghai Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJYY200907001
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2009-09

CONDITIONS: Chemoradiotherapy
Keywords: Intensity Modulated Radiation Therapy; Capecitabine; Resectable Rectal Carcinoma
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Preoperative Chemoradiotherapy — Patient will receive pre-operative radiotherapy with intensity modulated radiotherapy to primary and any grossly enlarged pelvic nodes 5Gy in 5 fractions over 5 days with concurrent capecitabine 1500mg p.o. bid for 1 week, then undergo surgery.
  Other Names: Capecitabine (Xeloda®)

SUMMARY:
Intensity modulated radiotherapy (IMRT)-based radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Investigators initiated a prospective study to evaluate the efficacy and toxicity of short course preoperative chemoradiotherapy utilizing Intensity Modulated Radiation Therapy (IMRT) in combination with capecitabine in patients with resectable rectal carcinoma.

DETAILED DESCRIPTION:
Preoperative chemoradiotherapy has become a standard part of treatment protocols in stage II and III rectal cancer. Compared to postoperative chemoradiotherapy, the advantage of preoperative application of chemotherapeutics and irradiation includes improved compliance, reduced toxicity, and downstaging of the tumor in a substantial number of patients. The latter may enhance the rate of curative surgery, permit sphincter preservation in patients with low-sited tumors, and have a positive impact on the quality of life of these patients (Sauer et al, 2004).

The most widely used chemotherapeutic agent in colorectal cancer has been 5-fluorouracil (5-FU), and numerous attempts have been made to improve its efficacy, including biomodulation and protracted infusion. It has been demonstrated that biomodulation with leucovorin or levamisole was not effective in rectal cancer (Tepper et al, 2002), and protracted infusion of 5-FU was superior to bolus injection (O'Connell et al, 1994). New oral chemotherapeutic agents including capecitabine have been introduced and tried in colorectal cancer. Capecitabine is a tumor-selective fluoropyrimidine carbamate designed to achieve a higher intratumoral 5-FU level with lower systemic toxicity than intravenous administration of 5-FU (Shimma et al, 2000). It passes intact through the intestinal mucosa and is converted to 5-FU, preferentially in tumor tissue by thymidine phosphorylase (Schuller et al, 2000 ; Ishikawa et al, 1998 ; Miwa et al, 1998). Theoretically, oral capecitabine mimics the effect of protracted infusion of 5-FU without complications accompanying intravenous delivery (Liu et al, 1997). Moreover, experimental data using human cancer xenografts demonstrated up-regulation of thymidine phosphorylase by radiation (Sawada et al, 1999), constituting a synergistic effect. In two randomized Phase III trials, capecitabine showed a superior overall response rate and safety profile compared with 5-FU/lecovorinin for metastatic colorectal cancer (Van Cutsem et al, 2001; Hoff et al, 2001; Twelves, 2002). Intensity modulated radiotherapy (IMRT)-based radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. (Ballonoff et al, 2008)

With such encouraging outcomes, investigators initiated a prospective study to evaluate the efficacy and toxicity of short course preoperative chemoradiotherapy utilizing Intensity Modulated Radiation Therapy (IMRT) in combination with capecitabine in patients with resectable rectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of adenocarcinoma of the rectum by biopsy technique that does not completely excise the lesion (e.g., fine needle aspiration, core needle biopsy)
* Located up to 15 cm from the anal verge with no extension of malignant disease into the anal canal
* Stage IIIB-IIIC disease (T3-T4, N0-2, M0)(i.e., without evidence of distant metastases) tumor as determined by the following assessments:Colonoscopy and biopsy within the past 8 weeks; History/physical examination (including medication history screen for contraindications) within the past 8 weeks; Contrast-enhanced imaging of the abdomen and pelvis either by CT, MRI, or PET-CT (whole body preferred) within the past 8 weeks
* Chest x-ray (or CT) of the chest within the past 8 weeks to exclude distant metastases (except for patients who have had whole body PET-CT)
* Transrectal ultrasound (TRUS) within the past 8 weeks required to establish tumor stage
* TRUS not required if clinical exam, CT of the pelvis, and/or MRI demonstrates T4 lesion
* No synchronous primary colon carcinoma
* No evidence of distant metastases (M1)
* ANC ≥ 1,800/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention to achieve hemoglobin ≥ 8.0 g/dL allowed)
* AST < 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior invasive malignancy except nonmelanoma skin cancer unless disease free for a minimum of 3 years

Exclusion Criteria:

* Severe, active comorbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the past 12 months
* Transmural myocardial infarction within the past 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 30 days
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* AIDS
* Evidence of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake
* Known, existing uncontrolled coagulopathy, unless clinically stable on anticoagulation therapy for ≥ 2 weeks
* Evidence of peripheral neuropathy ≥ grade 2
* Prior allergic reaction to capecitabine
* Lack of physical integrity of the gastrointestinal tract (i.e., severe Crohn disease that results in malabsorption; significant bowel resection that would make one concerned about the absorption of capecitabine) or malabsorption syndrome that would preclude feasibility of oral chemotherapy (i.e., capecitabine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate if downstaging of tumor is observed after preoperative chemoradiotherapy: pathological T stage of disease in surgical specimen will be compared with preoperative T stage. | Every 21 days

SECONDARY OUTCOMES:
To evaluate survival after preoperative chemoradiotherapy. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Cao, MD, Principal Investigator — Ruijin Hospital; Ren Zhao, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Department of General Surgery, Shanghai Ruijin Hospital, Shanghai
  - Department of Oncology, Shanghai Ruijin Hospital, Shanghai